CLINICAL TRIAL: NCT02570373
Title: Phase 1, Open-label, Single-dose Study to Characterize the Elimination of Guselkumab Glycoform Variants in Healthy Subjects
Brief Title: A Study to Characterize the Elimination of Guselkumab Glycoform Variants in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR107879; CNTO1959NAP1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-09-16; First posted 2015-10-07 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy; Guselkumab
MeSH Terms: interventions — guselkumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Guselkumab (Experimental): Participant will receive a single intravenous (IV) infusion of guselkumab at a dose of 10 milligram per kilogram (mg/kg) over 60 minutes on Day 1.
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Guselkumab — Participant will receive a single intravenous (IV) infusion of guselkumab at a dose of 10 milligram per kilogram (mg/kg) over 60 minutes on Day 1.

SUMMARY:
The purpose of this study is to characterize the elimination of guselkumab glycoform variants following a single intravenous (IV) administration of guselkumab at a 10 milligram per kilogram (mg/kg) dose in healthy participants.

DETAILED DESCRIPTION:
This is an open-label single-dose study in healthy participants. All participants will receive a single intravenous (IV) infusion of guselkumab at a dose of 10 milligram per kilogram (mg/kg) over 60 minutes on Day 1. After the administration of study drug on Day 1, participants will stay in the clinical study unit until being discharged after the assessments on Day 2. Participants will be required to return to the study center for outpatient visits including safety assessments through Day 85 after study drug administration. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be a healthy man or woman with no clinically significant abnormalities on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at Screening
* Participants must be otherwise healthy on the basis of clinical laboratory tests performed at Screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the subject may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Have a weight in the range of 60.0 kilogram (kg) to 100.0 kg, inclusive, if male; have a weight in the range of 50.0 kg to 90.0 kg, inclusive, if female. Have a body mass index of 18.5 kilogram per meter^2 (kg/m^2) to 30.0 kg/m^2, inclusive
* A woman must have a negative serum (beta human chorionic gonadotropin [beta hCG]) test at Screening and on Day -1
* Before drug administration, a woman must be either not of childbearing potential (Not of childbearing potential: Premenarchal; postmenopausal (greater than 45 years of age with amenorrhea for at least 12 months, or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) level > 40 international Units/ Liter); permanently sterilized (eg, tubal occlusion, hysterectomy, bilateral salpingectomy); or otherwise be incapable of pregnancy) OR of childbearing potential and practicing a highly effective method of birth control consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies (established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device (IUD) or intrauterine system (IUS); barrier methods: condom with spermicidal foam/gel/film/cream/suppository or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository; male partner sterilization (the vasectomized partner should be the sole partner for that participant); true abstinence [when this is in line with the preferred and usual lifestyle of the participant])

Exclusion Criteria:

* Participant currently has or has a history of any clinically significant medical illness or medical disorders the investigator considers should exclude the subject, including (but not limited to), neuromuscular, hematological disease, immune deficiency state, respiratory disease, hepatic or gastrointestinal (GI) disease, neurological or psychiatric disease, ophthalmological disorders, neoplastic disease, renal or urinary tract diseases, or dermatological disease
* Participant is currently undergoing or has previously undergone allergy immunotherapy for a history of anaphylactic reactions
* Participant has had major surgery (eg, requiring general anesthesia) within 8 weeks before screening, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study (16 weeks)
* Participant has previously received guselkumab
* Participant has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 3 months or 5 half-lives (whichever is longer) before the study drug administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-09-25 (Actual); Primary Completion 2016-01-12 (Actual); Study Completion 2016-01-12 (Actual)

PRIMARY OUTCOMES:
Change in Rate of Elimination of Guselkumab Glycoform Variants Following a Single IV Administration of Guselkumab at a 10 mg/kg Dose in Healthy Participants | Up to 43 days
  The composition of the glycoforms will be quantified and evaluated over time.

SECONDARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) as a Measure of Safety and Tolerability of CNTO1959 | up to 85 days
  Participant incidence of treatment-emergent adverse events, vital signs, physical examinations, laboratory safety tests, and 12-lead electrocardiograms (ECG).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Tempe, Arizona, United States

REFERENCES:
- See also: Phase 1, Open-label, Single-dose Study to Characterize the Elimination of Guselkumab Glycoform Variants in Healthy Subjects — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR107879&attachmentIdentifier=31c0c9f8-7e06-4239-ae92-4ab2bc6586a1&fileName=CR107879_CSR_Synopsis.pdf&versionIdentifier=